CLINICAL TRIAL: NCT01237418
Title: French Registry of Acute Coronary Syndrome With or Without ST Elevation 2010
Acronym: FAST-MI 2010
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 10240
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When normal blood test done at the patient's admission into ISB, an additional quantity of 60 ml of blood will be drawn up for building a DNAthèque (15 ml) and a serum bank (45 ml) on only markers related to atherosclerotic disease
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Myocardial Infarction: Any patient over 18 years admitted for myocardial infarction (MI) of less than 48 hours, characterized by the typical rise and fall of troponin or CPKMb

SUMMARY:
The observatory FAST MI 2010 proposes to establish a cohort of 3500 patients recruited prospectively over a period of 2 months.

Patients will be followed up at 1 month and then followed annually for 10 years.

Patients should have agreed to participate in the study, participation in the protocol, or refusal to participate will not affect the therapeutic approach of the physician. The study of genotypic or phenotypic characteristics will not change the therapeutic approach of health care teams.

DETAILED DESCRIPTION:
This is a multicenter observational study, given to 300 prospective medical facilities, CHU, CHG, CHR, health facility of the Army, including a clinic or intensive care unit entitled to receive emergency ACS. (See attached list 10-6) A questionnaire will be sent to each center before the recruitment center on the type and number of beds (Appendix 10-5)

Patients will be recruited consecutively in the CIAU member during a period of 2 months.

The 1-month follow-up will be done by the referring physician of each ISB, by mail or telephone contact with the treating physician and / or patient.

Annual follow-ups will be conducted during 10 years of clinical research technicians of the French Society of Cardiology, mail and / or telephone contact with the municipalities of birth, treating physicians and patients.

ELIGIBILITY:
Inclusion Criteria :

* Patients over 18 years old
* Admitted patient for a myocardial infarction (MI) of less than 48 hours, characterized by the typical rise and fall of troponin or CPKMb associated with at least one of the following: symptoms of myocardial ischemia or appearance of pathological Q waves or repolarization disorders related to ischemia (in addition to or NSTEMI)
* Patient who consented to participate in the study

Exclusion Criteria:

* Refusal of consent
* MI occurring within 48 h after a therapeutic intervention (angioplasty or coronary bypass or other surgery)
* Diagnosis of SCA reversed in favor of an alternative diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively in the CIAU member during a period of 2 months, including sub-populations of specific interest (diabetes and / or elderly patients, for example). A list of eligible patients not included and must be completed by the participating centers during the same period, with reasons for non inclusion.
  A questionnaire will be sent to each center prior to recruitment, including type of service and number of beds in the facility.
  The study will be given to any medical facility, University Hospital, CHG, CHR, health facility of the Army, including a clinic or intensive care unit entitled to receive emergency ACS. In each center, a medical consultant will be appointed to collect phenotypic data for the study case report forms in electronic patient.
Sampling Method: Probability Sample
Enrollment: 4168 (Actual)
Dates: Start 2010-10; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 1 month
  Compare survival in the hospital after admission in Intensive Care Unit in the manner of care

SECONDARY OUTCOMES:
Survival in long-term | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Danchin, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- European Hospital Georges Pompidou, Paris, France

REFERENCES:
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Danchin N, Fauchier L, Marijon E, Barnay C, Furber A, Mabo P, Bernard P, Blanc JJ, Jouven X, Le Heuzey JY, Charbonnier B, Ferrieres J, Simon T; French registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction (FAST-MI) Investigators. Impact of early statin therapy on development of atrial fibrillation at the acute stage of myocardial infarction: data from the FAST-MI register. Heart. 2010 Nov;96(22):1809-14. doi: 10.1136/hrt.2010.201574. PMID 20965993
- [Background] Zeller M, Danchin N, Simon D, Vahanian A, Lorgis L, Cottin Y, Berland J, Gueret P, Wyart P, Deturck R, Tabone X, Machecourt J, Leclercq F, Drouet E, Mulak G, Bataille V, Cambou JP, Ferrieres J, Simon T; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction investigators. Impact of type of preadmission sulfonylureas on mortality and cardiovascular outcomes in diabetic patients with acute myocardial infarction. J Clin Endocrinol Metab. 2010 Nov;95(11):4993-5002. doi: 10.1210/jc.2010-0449. Epub 2010 Aug 11. PMID 20702526
- [Background] Danchin N, Coste P, Ferrieres J, Steg PG, Cottin Y, Blanchard D, Belle L, Ritz B, Kirkorian G, Angioi M, Sans P, Charbonnier B, Eltchaninoff H, Gueret P, Khalife K, Asseman P, Puel J, Goldstein P, Cambou JP, Simon T; FAST-MI Investigators. Comparison of thrombolysis followed by broad use of percutaneous coronary intervention with primary percutaneous coronary intervention for ST-segment-elevation acute myocardial infarction: data from the french registry on acute ST-elevation myocardial infarction (FAST-MI). Circulation. 2008 Jul 15;118(3):268-76. doi: 10.1161/CIRCULATIONAHA.107.762765. Epub 2008 Jun 30. PMID 18591434
- [Result] Hanssen M, Cottin Y, Khalife K, Hammer L, Goldstein P, Puymirat E, Mulak G, Drouet E, Pace B, Schultz E, Bataille V, Ferrieres J, Simon T, Danchin N; FAST-MI 2010 Investigators. French Registry on Acute ST-elevation and non ST-elevation Myocardial Infarction 2010. FAST-MI 2010. Heart. 2012 May;98(9):699-705. doi: 10.1136/heartjnl-2012-301700. PMID 22523054
- [Result] Puymirat E, Aissaoui N, Simon T, Bataille V, Drouet E, Mulak G, Ferrieres J, Danchin N. [Acute myocardial infarction in the elderly. The FAST-MI registry]. Presse Med. 2013 Nov;42(11):1432-41. doi: 10.1016/j.lpm.2013.04.010. Epub 2013 Jul 22. French. PMID 23886929
- [Result] Simon T, Puymirat E, Lucke V, Bouabdallaoui N, Lognone T, Aissaoui N, Cohen S, Ashrafpoor G, Roul G, Jouve B, Levy G, Charpentier S, Grollier G, Ferrieres J, Danchin N; au nom des investigateurs FAST-MI 2010. [Acute myocardial infarction in women. Initial characteristics, management and early outcome. The FAST-MI registry]. Ann Cardiol Angeiol (Paris). 2013 Aug;62(4):221-6. doi: 10.1016/j.ancard.2013.06.003. Epub 2013 Jul 4. French. PMID 23920136
- [Result] Puymirat E, Teixeira N, Simon T, Steg PG, Schiele F, Lamblin N, Probst V, Juilliere Y, Ferrieres J, Danchin N; FAST-MI investigators. Patient education after acute myocardial infarction: cardiologists should adapt their message--French registry of acute ST-elevation or non-ST-elevation myocardial infarction 2010 registry. J Cardiovasc Med (Hagerstown). 2015 Nov;16(11):761-7. doi: 10.2459/JCM.0000000000000092. PMID 24751516
- [Result] Puymirat E, Schiele F, Ennezat PV, Coste P, Collet JP, Bonnefoy-Cudraz E, Roul G, Richard P, Simon T, Danchin N. Impact of fondaparinux versus enoxaparin on in-hospital bleeding and 1-year death in non-ST-segment elevation myocardial infarction. FAST-MI (French Registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction) 2010. Eur Heart J Acute Cardiovasc Care. 2015 Jun;4(3):211-9. doi: 10.1177/2048872614544857. Epub 2014 Jul 29. PMID 25075006
- [Result] Puymirat E, Aissaoui N, Cottin Y, Vanzetto G, Carrie D, Isaaz K, Valy Y, Tchetche D, Schiele F, Steg PG, Simon T, Danchin N. Effect of coronary thrombus aspiration during primary percutaneous coronary intervention on one-year survival (from the FAST-MI 2010 registry). Am J Cardiol. 2014 Dec 1;114(11):1651-7. doi: 10.1016/j.amjcard.2014.08.039. Epub 2014 Sep 16. PMID 25304976
- [Result] Puymirat E, Schiele F, Steg PG, Blanchard D, Isorni MA, Silvain J, Goldstein P, Gueret P, Mulak G, Berard L, Bataille V, Cattan S, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Determinants of improved one-year survival in non-ST-segment elevation myocardial infarction patients: insights from the French FAST-MI program over 15 years. Int J Cardiol. 2014 Nov 15;177(1):281-6. doi: 10.1016/j.ijcard.2014.09.023. Epub 2014 Sep 28. PMID 25499393
- [Result] Puymirat E, Caudron J, Steg PG, Lemesle G, Cottin Y, Coste P, Schiele F, de Labriolle A, Bataille V, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Prognostic impact of non-compliance with guidelines-recommended times to reperfusion therapy in ST-elevation myocardial infarction. The FAST-MI 2010 registry. Eur Heart J Acute Cardiovasc Care. 2017 Feb;6(1):26-33. doi: 10.1177/2048872615610893. Epub 2016 Sep 20. PMID 26450784
- [Result] Bailleul C, Puymirat E, Aissaoui N, Schiele F, Ducrocq G, Coste P, Blanchard D, Brasselet C, Elbaz M, Steg PG, Le Breton H, Bonnefoy-Cudraz E, Montalescot G, Cottin Y, Goldstein P, Ferrieres J, Simon T, Danchin N; FAST-MI Investigators. Factors Associated With Infarct-Related Artery Patency Before Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction (from the FAST-MI 2010 Registry). Am J Cardiol. 2016 Jan 1;117(1):17-21. doi: 10.1016/j.amjcard.2015.09.043. Epub 2015 Oct 23. PMID 26541905
- [Result] Sokoloff A, Lefevre G, Teixeira N, Puymirat E, Beygui F, Vanzetto G, Richard P, Khalife K, Blanchard D, Gilard M, Coste P, Farah B, Elbaz M, Leclercq F, Ferrari E, Bonnet JL, Meyer P, Belle L, Funck F, Motreff P, Virot P, Geugniaud PY, Ferrieres J, Simon T, Danchin N. [Characteristics and management of ST-elevation myocardial infarction in France: Regional variations in 2010]. Ann Cardiol Angeiol (Paris). 2015 Dec;64(6):427-33. doi: 10.1016/j.ancard.2015.10.001. Epub 2015 Nov 5. French. PMID 26547524
- [Result] Puymirat E, Lamhaut L, Bonnet N, Aissaoui N, Henry P, Cayla G, Cattan S, Steg G, Mock L, Ducrocq G, Goldstein P, Schiele F, Bonnefoy-Cudraz E, Simon T, Danchin N. Correlates of pre-hospital morphine use in ST-elevation myocardial infarction patients and its association with in-hospital outcomes and long-term mortality: the FAST-MI (French Registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction) programme. Eur Heart J. 2016 Apr 1;37(13):1063-71. doi: 10.1093/eurheartj/ehv567. Epub 2015 Nov 17. PMID 26578201
- [Result] Massoullie G, Wintzer-Wehekind J, Chenaf C, Mulliez A, Pereira B, Authier N, Eschalier A, Clerfond G, Souteyrand G, Tabassome S, Danchin N, Citron B, Lusson JR, Puymirat E, Motreff P, Eschalier R. Prognosis and management of myocardial infarction: Comparisons between the French FAST-MI 2010 registry and the French public health database. Arch Cardiovasc Dis. 2016 May;109(5):303-10. doi: 10.1016/j.acvd.2016.01.012. Epub 2016 Apr 20. PMID 27107986
- [Result] Schiele F, Puymirat E, Bonello L, Meneveau N, Collet JP, Motreff P, Ravan R, Leclercq F, Ennezat PV, Ferrieres J, Simon T, Danchin N. Switching between thienopyridines in patients with acute myocardial infarction and quality of care. Open Heart. 2016 May 23;3(1):e000384. doi: 10.1136/openhrt-2015-000384. eCollection 2016. PMID 27252877
- [Result] Aissaoui N, Puymirat E, Juilliere Y, Jourdain P, Blanchard D, Schiele F, Gueret P, Popovic B, Ferrieres J, Simon T, Danchin N. Fifteen-year trends in the management of cardiogenic shock and associated 1-year mortality in elderly patients with acute myocardial infarction: the FAST-MI programme. Eur J Heart Fail. 2016 Sep;18(9):1144-52. doi: 10.1002/ejhf.585. PMID 27594176
- [Result] Puymirat E, Aissaoui N, Lemesle G, Cottin Y, Coste P, Schiele F, Ferrieres J, Simon T, Danchin N; FAST-MI Investigators. Long-Term Clinical Outcomes According to Previous Manifestations of Atherosclerotic Disease (from the FAST-MI 2010 Registry). Am J Cardiol. 2017 Mar 1;119(5):692-697. doi: 10.1016/j.amjcard.2016.11.032. Epub 2016 Dec 2. PMID 28038725
- [Result] Puymirat E, Aissaoui N, Cayla G, Lafont A, Riant E, Mennuni M, Saint-Jean O, Blanchard D, Jourdain P, Elbaz M, Henry P, Bataille V, Drouet E, Mulak G, Schiele F, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Changes in One-Year Mortality in Elderly Patients Admitted with Acute Myocardial Infarction in Relation with Early Management. Am J Med. 2017 May;130(5):555-563. doi: 10.1016/j.amjmed.2016.12.005. Epub 2017 Jan 5. PMID 28065766
- [Result] Schiele F, Gale CP, Simon T, Fox KAA, Bueno H, Lettino M, Tubaro M, Puymirat E, Ferrieres J, Meneveau N, Danchin N. Assessment of Quality Indicators for Acute Myocardial Infarction in the FAST-MI (French Registry of Acute ST-Elevation or Non-ST-Elevation Myocardial Infarction) Registries. Circ Cardiovasc Qual Outcomes. 2017 Jun;10(6):e003336. doi: 10.1161/CIRCOUTCOMES.116.003336. PMID 28630371
- [Result] Puymirat E, Simon T, Cayla G, Cottin Y, Elbaz M, Coste P, Lemesle G, Motreff P, Popovic B, Khalife K, Labeque JN, Perret T, Le Ray C, Orion L, Jouve B, Blanchard D, Peycher P, Silvain J, Steg PG, Goldstein P, Gueret P, Belle L, Aissaoui N, Ferrieres J, Schiele F, Danchin N; USIK, USIC 2000, and FAST-MI investigators. Acute Myocardial Infarction: Changes in Patient Characteristics, Management, and 6-Month Outcomes Over a Period of 20 Years in the FAST-MI Program (French Registry of Acute ST-Elevation or Non-ST-Elevation Myocardial Infarction) 1995 to 2015. Circulation. 2017 Nov 14;136(20):1908-1919. doi: 10.1161/CIRCULATIONAHA.117.030798. Epub 2017 Aug 27. PMID 28844989
- [Result] Bailleul C, Aissaoui N, Cayla G, Dillinger JG, Jouve B, Schiele F, Ferrieres J, Simon T, Danchin N, Puymirat E; FAST-MI investigators. Prognostic impact of prepercutaneous coronary intervention TIMI flow in patients with ST-segment and non-ST-segment elevation myocardial infarction: Results from the FAST-MI 2010 registry. Arch Cardiovasc Dis. 2018 Feb;111(2):101-108. doi: 10.1016/j.acvd.2017.04.004. Epub 2017 Sep 19. PMID 28939193
- [Result] Puymirat E, Aissaoui N, Bonello L, Cayla G, Labeque JN, Nallet O, Motreff P, Varenne O, Schiele F, Ferrieres J, Simon T, Danchin N; FAST-MI Investigators. Clinical outcomes according to symptom presentation in patients with acute myocardial infarction: Results from the FAST-MI 2010 registry. Clin Cardiol. 2017 Dec;40(12):1256-1263. doi: 10.1002/clc.22819. Epub 2017 Dec 15. PMID 29243857
- [Result] Aissaoui N, Riant E, Lefevre G, Delmas C, Bonello L, Henry P, Bonnefoy E, Schiele F, Ferrieres J, Simon T, Danchin N, Puymirat E; FAST-MI investigators. Long-term clinical outcomes in patients with cardiogenic shock according to left ventricular function: The French registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction (FAST-MI) programme. Arch Cardiovasc Dis. 2018 Nov;111(11):678-685. doi: 10.1016/j.acvd.2017.11.002. Epub 2017 Dec 28. PMID 29290598
- [Result] Isorni MA, Aissaoui N, Angoulvant D, Bonello L, Lemesle G, Delmas C, Henry P, Schiele F, Ferrieres J, Simon T, Danchin N, Puymirat E; FAST-MI investigators. Temporal trends in clinical characteristics and management according to sex in patients with cardiogenic shock after acute myocardial infarction: The FAST-MI programme. Arch Cardiovasc Dis. 2018 Oct;111(10):555-563. doi: 10.1016/j.acvd.2018.01.002. Epub 2018 Feb 22. PMID 29478810
- [Result] Puymirat E, Simon T, Danchin N; FAST-MI Investigators. Response by Puymirat et al to Letter Regarding Article, "Acute Myocardial Infarction Changes in Patient Characteristics, Management, and 6-Month Outcomes Over a Period of 20 Years in the FAST-MI Program (French Registry of Acute ST Elevation or Non-ST-Elevation Myocardial Infarction) 1995 to 2015". Circulation. 2018 May 22;137(21):2307-2308. doi: 10.1161/CIRCULATIONAHA.118.033969. No abstract available. PMID 29784688
- [Result] Puymirat E, Cayla G, Cottin Y, Elbaz M, Henry P, Gerbaud E, Lemesle G, Popovic B, Labeque JN, Roubille F, Andrieu S, Farah B, Schiele F, Ferrieres J, Simon T, Danchin N. Twenty-year trends in profile, management and outcomes of patients with ST-segment elevation myocardial infarction according to use of reperfusion therapy: Data from the FAST-MI program 1995-2015. Am Heart J. 2019 Aug;214:97-106. doi: 10.1016/j.ahj.2019.05.007. Epub 2019 May 16. PMID 31181374
- [Result] Schiele F, Puymirat E, Ferrieres J, Simon T, Fox KAA, Eikelboom J, Danchin N; FAST-MI investigators. The FAST-MI 2005-2010-2015 registries in the light of the COMPASS trial: The COMPASS criteria applied to a post-MI population. Int J Cardiol. 2019 Mar 1;278:7-13. doi: 10.1016/j.ijcard.2018.11.138. Epub 2018 Dec 3. PMID 30538057
- [Result] Tea V, Bonaca M, Chamandi C, Iliou MC, Lhermusier T, Aissaoui N, Cayla G, Angoulvant D, Ferrieres J, Schiele F, Simon T, Danchin N, Puymirat E; FAST-MI investigators. Appropriate secondary prevention and clinical outcomes after acute myocardial infarction according to atherothrombotic risk stratification: The FAST-MI 2010 registry. Eur J Prev Cardiol. 2019 Mar;26(4):411-419. doi: 10.1177/2047487318808638. Epub 2018 Oct 24. PMID 30354737
- [Result] Puymirat E, Bonaca M, Iliou MC, Tea V, Ducrocq G, Douard H, Labrunee M, Plastaras P, Chevallereau P, Taldir G, Bataille V, Ferrieres J, Schiele F, Simon T, Danchin N; FAST-MI investigators. Outcome associated with prescription of cardiac rehabilitation according to predicted risk after acute myocardial infarction: Insights from the FAST-MI registries. Arch Cardiovasc Dis. 2019 Aug-Sep;112(8-9):459-468. doi: 10.1016/j.acvd.2019.04.002. Epub 2019 May 22. PMID 31126738
- [Result] Puymirat E, Bonaca M, Fumery M, Tea V, Aissaoui N, Lemesles G, Bonello L, Ducrocq G, Cayla G, Ferrieres J, Schiele F, Simon T, Danchin N; FAST-MI investigators. Atherothrombotic risk stratification after acute myocardial infarction: The Thrombolysis in Myocardial Infarction Risk Score for Secondary Prevention in the light of the French Registry of Acute ST Elevation or non-ST Elevation Myocardial Infarction registries. Clin Cardiol. 2019 Feb;42(2):227-234. doi: 10.1002/clc.23131. Epub 2018 Dec 27. PMID 30536449
- [Result] Ferrieres J, Bataille V, Puymirat E, Schiele F, Simon T, Danchin N; FAST-MI investigators. Applicability of the REDUCE-IT trial to the FAST-MI registry. Are the results of randomized trials relevant in routine clinical practice? Clin Cardiol. 2020 Nov;43(11):1260-1265. doi: 10.1002/clc.23437. Epub 2020 Jul 28. PMID 32720384
- [Derived] Fayol A, Schiele F, Ferrieres J, Puymirat E, Bataille V, Tea V, Chamandi C, Albert F, Lemesle G, Cayla G, Weizman O, Simon T, Danchin N; FAST-MI Investigators. Association of Use and Dose of Lipid-Lowering Therapy Post Acute Myocardial Infarction With 5-Year Survival in Older Adults. Circ Cardiovasc Qual Outcomes. 2024 May;17(5):e010685. doi: 10.1161/CIRCOUTCOMES.123.010685. Epub 2024 Apr 29. PMID 38682335
- [Derived] Garcia R, Marijon E, Karam N, Narayanan K, Anselme F, Cesari O, Champ-Rigot L, Manenti V, Martins R, Puymirat E, Ferrieres J, Schiele F, Simon T, Danchin N. Ventricular fibrillation in acute myocardial infarction: 20-year trends in the FAST-MI study. Eur Heart J. 2022 Dec 14;43(47):4887-4896. doi: 10.1093/eurheartj/ehac579. PMID 36303402
- [Derived] Dillinger JG, Achkouty G, Albert F, Muller G, Labeque JN, Moisson L, Morelle JF, Cottin Y, Pezel T, Lim P, Aissaoui N, Schiele F, Ferrieres J, Angoulvant D, Henry P, Puymirat E, Simon T, Danchin N; FAST-MI investigators. Deleterious synergistic effects of acute heart failure and diabetes mellitus in patients with acute coronary syndrome: Data from the FAST-MI Registries. Arch Cardiovasc Dis. 2022 May;115(5):264-275. doi: 10.1016/j.acvd.2022.02.004. Epub 2022 Mar 4. PMID 35304066
- [Derived] Danchin N, Puymirat E, Cayla G, Cottin Y, Coste P, Gilard M, Goldstein P, Braun F, Belle L, Montalescot G, Ferrieres J, Schiele F, Simon T; FAST-MI Investigators. One-Year Survival After ST-Segment-Elevation Myocardial Infarction in Relation With Prehospital Administration of Dual Antiplatelet Therapy. Circ Cardiovasc Interv. 2018 Sep;11(9):e007241. doi: 10.1161/CIRCINTERVENTIONS.118.007241. PMID 30354592